CLINICAL TRIAL: NCT06827249
Title: A Multicenter, Randomized, Positive-controlled, Non-inferiority Clinical Study to Evaluate the Safety and Efficacy of Peginterferon α2b Injection in the Treatment of Pediatric RSV Bronchiolitis
Brief Title: Peginterferon α-2b Injection for the Treatment of Pediatric RSV Bronchiolitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Hao Chuangli, Chief physician, Children's Hospital of Soochow University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Peg IFN α- 2b and atomization
Record Dates: First submitted 2025-01-21; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Peginterferon α-2b; respiratory syncytial virus
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peginterferon α-2b 90 mcg dose group (Experimental): The experimental group participants inhaled Peginterferon on the basis of receiving symptomatic supportive treatment.
  Interventions: Drug: Peginterferon α-2b injection
- Recombinant human interferon α-2b dose group (Active Comparator): The control group participants received symptomatic supportive treatment and aerosolized inhalation therapy with recombinant human interferon α-2b.
  Interventions: Drug: Recombinant Human Interferon α2b

INTERVENTIONS:
Drug: Peginterferon α-2b injection — Peginterferon α-2b injection, 90 mcg, on the basis of conventional treatments such as asthma control, oxygen inhalation, and fluid replacement, nebulized inhalation using air compression or oxygen-driven methods is administered on days 1, 3, and 5, once a day.
  Arms: Peginterferon α-2b 90 mcg dose group
Drug: Recombinant Human Interferon α2b — Recombinant Human Interferon alpha 2b, at a dose of 100,000 IU/kg, based on the conventional treatments such as asthma control, oxygen inhalation, and fluid replacement, will be administered via nebulized inhalation using air compression or oxygen-driven methods from day 1 to day 5, twice daily.
  Arms: Recombinant human interferon α-2b dose group

SUMMARY:
This is a multicenter, randomized, positive-controlled, non-inferiority clinical study, planning to enroll 90 children with bronchiolitis caused by respiratory syncytial virus infection, to evaluate the safety and efficacy of inhaled Peginterferon α-2b injection compared to recombinant human interferon α2b in the treatment of pediatric respiratory syncytial virus bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

1. The guardian of the child is able to understand the content, requirements, and limitations of the protocol, fully understands the possible adverse reactions that may occur during the study, is willing to complete the follow-up as required, and voluntarily signs the informed consent form before the start of the study.
2. The child's age is 6 months or older but no more than 2 years old (including the critical value) at the time of signing the informed consent, and the gender is not specified.
3. Positive viral detection in nasopharyngeal swab.
4. Presence of rapid breathing, wheezing, moist rales and/or wheezing sounds in the lungs; with or without chest imaging showing signs of hyperinflation, patchy infiltrates, localized atelectasis, and peribronchitis.
5. The severity of the illness is mild or moderate (evaluation criteria see Appendix 1: Wang Bronchiolitis Scoring Standard).
6. The time from the onset of the child's illness to the signing of the informed consent form is within 72 hours (the appearance of symptoms and signs related to RSV bronchiolitis does not exceed 72 hours from the signing of the informed consent, including but not limited to: tachypnea, wheezing, hypoxemia, dyspnea, fever).
7. No use of other antiviral drugs or immunomodulators within 3 weeks before randomization.

Exclusion Criteria:

1. Extreme restlessness, drowsiness, coma, and possibly requiring mechanical ventilation assistance for breathing.
2. Presence of other chronic severe diseases such as cardiac insufficiency, respiratory insufficiency, liver insufficiency, renal insufficiency, and severe malnutrition.
3. Having autoimmune diseases such as systemic lupus erythematosus or psoriasis, or immunodeficiency diseases.
4. Having epilepsy or other disorders of central nervous system function.
5. The investigator's comprehensive judgment suspects a concurrent bacterial infection.
6. Clinical diagnosis of myocarditis or suspected myocarditis (diagnostic criteria see Appendix 2: Diagnostic Recommendations for Myocarditis in Children).
7. Known or suspected allergy to interferon or excipients.
8. Participation in other interventional clinical trials within 3 months prior to screening, or planning to participate in other clinical trials during the study period. (9) A history of pneumonia in the past 3 months.

(10) Other conditions deemed unsuitable for inclusion by the investigator.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The rate of change in Wang's bronchiolitis score from baseline. | Day 6.

SECONDARY OUTCOMES:
Wang's bronchiolitis score change from baseline. | Day1-7.
The proportion of Wang's bronchiolitis score being 0 points. | Day6.
Length of hospital stay. | through study completion, an average of 18 months
Duration of oxygen therapy support. | through study completion, an average of 18 months
Change in viral load from baseline. | through study completion, an average of 18 months
Adverse Event(AE). | through study completion, an average of 18 months
Body temperature. | through study completion, an average of 18 months
Number of Participants with Abnormal Laboratory Parameters Findings. | through study completion, an average of 18 months
The number of research subjects who withdrew early. | through study completion, an average of 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Chuangli Hao, Ph.D, Principal Investigator — Children's Hospital of Soochow University; Fanzheng Meng, Ph.D, Study Director — The First Hospital of Jilin University; Xiaoxia Lu, Ph.D, Study Director — Wuhan women and children's health care center
Locations (3):
- China (3):
  - Wuhan Women and Children's Health Care Center, Wuhan, Hubei
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No